CLINICAL TRIAL: NCT06889324
Title: Efficacy of Vibration Therapy on Restless Legs Syndrome and Sleep Disturbances Among Patients Undergoing Hemodialysis
Acronym: RLS-Sleep
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amjed Abdulabbas Shraida (Other)
Responsible Party: Sponsor-Investigator, Amjed Abdulabbas Shraida, Lecturer, Kufa University
Organization: Kufa University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaghdadU
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Sleep disturbances; Hemodialysis
MeSH Terms: conditions — Restless Legs Syndrome; Parasomnias

STUDY DESIGN:
Intervention Model Description: Patients with legs restless syndrome and sleep disturbances during hemodialysis will be assessed for eligibility. After that, the researcher will use a simple random sampling technique by writing the names of the patients on slips of paper and placing them in a bowl, mixing them well, and then pulling them randomly to allocate them into two groups; half patients as a study group will take vibration therapy applied on the calf muscle for 10 minutes per session, 2 times per week for total one month, during the first hour of each hemodialysis sessions, and the other half patients will not exposed to the therapy and will take only routine care and considered as the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration therapy (Experimental): Experimental group will take vibration therapy applied on the calf muscle for 10 minutes per session, 2 times per week for total one month, during the first hour of each hemodialysis sessions
  Interventions: Other: Vibration therapy
- Routine care (No Intervention): Control group will not exposed to the vibration therapy and will take only routine care.

INTERVENTIONS:
Other: Vibration therapy — Its therapy uses mechanical vibrations delivered via a specialized device called Thrive vibrator device model 717 to stimulate the calf muscles, which can help reduce the severity of restless legs syndrome and sleep disturbances among patients undergoing hemodialysis.
  Arms: Vibration therapy

SUMMARY:
The goal of this clinical trial is to learn if whether vibration therapy relieves the intensity of Restless legs syndrome (RLS) symptoms and sleep disturbances among patients undergoing hemodialysis. The main question it aims to answer is:

Is there a difference in the levels of legs restless syndrome and sleep disturbances between hemodialysis patients who receive vibration therapy and those who do not receive it?

Researcher will compare the levels of legs restless syndrome and sleep disturbances between hemodialysis patients who receive vibration therapy and those who do not receive it to see if vibration therapy works to relieve the levels of legs restless syndrome and sleep disturbances.

Participants will take vibration therapy applied on the calf muscle for 10 minutes per session, 2 times per week for total one month, during the first hour of each hemodialysis sessions.

DETAILED DESCRIPTION:
Background Most hemodialysis patients are faced with a variety of complications such as restless leg syndrome and sleep disorders during the course of their disease. Restless legs syndrome (RLS) is one of the most prevalent problems in patients receiving hemodialysis. Studies indicate that the prevalence of this sensorimotor neurological disorder in hemodialysis patients ranges from (6.6%) to (80%), contrasted to (7%) to (24.1%) in the general population. RLS adversely affects outcomes of patients with chronic renal failure receiving long-term hemodialysis, with significant impacts on sleep quality and quality of life, as well as increased mortality after 2.5 years of follow-up.

In terms of sleep, the quality of sleep in hemodialysis patients is often affected by restless legs syndrome. The individual feels very disturbing, deep creeping sensations inside the leg whenever sitting or lying down. These abnormal sensations cause insomnia, daytime sleepiness, shorter sleep duration, and the use of sedatives and hypnotics. Sleep disturbances and deprivation of sleep induced by RLS can impact the sleep quality and emotional well-being of patients undergoing hemodialysis, potentially resulting in depression, anxiety, and increment risk of cardiovascular issues.

Dialysis nurses should manage hemodialysis problems using efficient nonpharmacological techniques. As previously said, RLS significantly effects on both the physical and mental soundness of patients, in addition to disrupting their daily lives. Furthermore, many of the medications used to treat these individuals are mostly eliminated by the kidneys, producing further complications for the patients. These matters underscore the need of employing non-pharmacological approaches to treat restless legs syndrome and sleep disorders.

Importance of study There are approximately 3,730,000 patients with Chronic kidney Disease (CKD) globally, and the annual growth rate of the disease is 5-6%. According to data, more than 2.5 million patients with end-stage kidney disease are currently undergoing renal replacement therapy (RRT), and this figure is expected to rise to around 4.5 million by 2030. For patients with CKD, the most prevalent technique of RRT is hemodialysis.

Patients with kidney failure receiving continuous hemodialysis experience a variety of symptoms, including restless leg syndrome (RLS) and sleep disturbances. RLS is a clinical disorder with a prevalence ranging from 6.6% to 83% among patients receiving hemodialysis. It is characterized by a strong desire to move the legs, and this desire usually take place in the afternoon and evening. The moving desire is accompanied by uncomfortable and frequently painful feelings in the legs. The legs movement can help reduce painful and uncomfortable legs feelings. Above 90% of individuals with RLS have periodic leg movements (PLM) during sleeping. The periodic leg movements (PLMs) are sporadic and cause involuntary foot dorsiflexion, knee flexion, and sometimes thigh flexion, occurring every 20 to 40 seconds. The uncomfortable nighttime sensibility and need to move the legs generate intermittent movements of leg during sleep, which lateness and disrupt sleep, resulting in repeated awakenings, and promoting daytime drowsiness, all of which reduce the quality of life for patients.

Regarding sleep, Sleep disorders are common issues that many patients on hemodialysis experience. It is thought that these individuals have a prevalence of sleep problems that varies from 18% to 69% in different forms, such as patients with restless leg syndrome linked to obstructive sleep apnea. Sleep quality refers to an individual's contentment with their sleep experience, which encompasses many aspects like how quickly fall asleep, the total duration of sleep, the ability to stay asleep, and the feeling of being refreshed upon waking. Deprivation of sleep produces many issues like chronic weariness, malfunction, alterations in the neurological system, and decreased willingness to care for oneself, thus it is essential to focus on sleep quality and address sleep deprivation in patients undergoing hemodialysis.

Many pharmacological or non-pharmacological therapies can be used to treat patients with end-stage renal disease (ESKD) who have restless legs syndrome (RLS) and sleep disturbances. RLS treatments include dopamine agonists (pramipexole and ropinirole), antiepileptics (gabapentin), hypnotics, opiates (tramadol), and sedatives. Despite their effectiveness in alleviating symptoms and improving sleep time, these drugs have side effects such as headache, general weakness, nausea, emesis, and drowsiness, which eventually cause the symptoms of RLS to rebound and worsen. As for non-pharmacological approach, which include many interventions such as vibration, massage, exercise, aromatherapy, reflexology, cryotherapy, and cold dialysis, they have been reported to reduce the symptoms of restless legs syndrome in patients receiving hemodialysis. Unfortunately, these non-pharmacological approaches are offered in randomized studies that lack well-determined control groups, leading to a loss of clarity in the objective analysis of the study results. In addition, Salib and others encourage further studies involving a larger patient population and longer follow-up periods to identify the most suitable, safe, and cost-effective methods for managing this condition in hemodialysis patients. Conducting a study fills this gap by providing empirical data to support or refute the potential benefits of this intervention. This contributes to the evidence base in nephrology and rehabilitation medicine.

So the current study aims to find out whether vibration therapy relieves the intensity of RLS symptoms and sleep disturbances among patients undergoing hemodialysis. Exploring how vibration therapy affects symptoms like RLS and sleep disturbances can provide insights into the underlying mechanisms of these conditions in hemodialysis patients. As well as the positive findings from the study could potentially influence clinical practice guidelines for managing RLS and sleep disturbances in hemodialysis settings. Healthcare providers may consider integrating vibration therapy into multidisciplinary treatment plans to enhance symptom management and improve patient outcomes.

Research design:

In the current study, the researcher will utilize a pretest-posttest randomized controlled trial design.

Setting:

The study will be conducted in Al-Najaf City/Al-Najaf Al-Ashraf Health Directorate / Al-Sadder Medical City / The Specialized Center for Kidney Diseases and Transplantation / Hemodialysis Unit. This center was chosen due to the availability of patients, in addition to the fact that patients undergo dialysis treatment according to a specific schedule, which helps researcher to control the follow-up of patients.

Study samples:

Patients undergoing hemodialysis who have legs restless syndrome and sleep disturbances.

Sampling method :

According to Consolidated Standards of Reporting Trials (CONSORT), the patients undergoing hemodialysis will be assessed for eligibility to assign the sample for the study. The sample will then be allocated randomly into two groups; the study group and the control group, in this step a simple random sampling technique well be used to ensure that selection is unbiased and every individual has an equal chance of being chosen in order to achieve randomization when the sample is allocated into two groups.

Minimum sample size:

The sample size for the current study will be established using the G-Power analysis approach. The G-Power analysis method includes three parameters; power (minimum 80%), significance (0.05), and effect size. The researcher identified the following determinants to determine the sample size in the current study with a power greater than (95%): Significance (0.05), and effect size (0.5). So, the required sample size equals 70 (35 study group and 35 control group).

Data analysis:

The following statistical data analysis technique will be utilized to examine the study's data using the IBM Statistical Package for Social Science (SPSS) Ver. (19) and Microsoft Excel (2010):

1. Descriptive Data Analysis:

   1. Tables (Frequencies, and Percentages).
   2. Statistical figures (Bar Charts).
   3. Statistical mean and standard deviation.
2. Inferential Data Analysis:

   1. Paired sample t-test to identifying the mean difference between the pre-test and post-test for the control group.
   2. ANOVA: To compare the difference in the mean values of levels of legs restless syndrome and sleep disturbances among the participants of study group throughout three periods of measurements.
   3. Regression: to determine the relationship between socio-demographic data with Post-test 1 and Post-test 2 for the study group.

ELIGIBILITY:
Inclusion Criteria:

* Patients passing at least three months after first their hemodialysis
* Patients who are receiving two or more HD sessions a week, to facilitate patient follow-up.
* Patients who are willing to participate, because the patients' participation is voluntary.
* Patients who are alert and able to communicate verbally, to make the program applicable and facilitate the data collection.

Exclusion Criteria:

* Emergency hemodialysis patients, to avoid mal-efficient (apply the program in a harmless manner).
* Intake of drugs for restless leg syndrome and sleep disturbances.
* Using vibration and massage therapy at home
* Recent history of deep vein thrombosis or other vascular complications.
* Patients who are unable to communicate, because the patients' communication is an essential part of data collection.
* Patients with severe cardiovascular disorders such as unstable angina, recent myocardial infarction or severe heart failure, because the application of the program may increase cardiovascular stress, which may pose a risk to these patients.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Arabic version of the Restless Legs Syndrome Rating Scale | There will be three time points at which the measurement is assessed for both the study and the control group as follows: Pre-test: At the first day Post-test 1: two weeks later . Post-test 2: four weeks later.
  A five-level Likert rating scale will be employed for rating the severity of Legs Restless Syndrome among patients receiving hemodialysis, ranging from (0 to 4) where (0) representing no RLS, (1) representing mild RLS, (2) representing moderate RLS, (3) representing severe RLS, and (4) represents very severe RLS. The scale consists of 10 items, and the maximum total score for the patient's answers is (40), higher scores indicate more severe symptoms. The severity of RLS is scored as (0) for no RLS, (1 - 10) for mild RLS, (11 - 20) for moderate RLS, (21 - 30) for severe RLS, and (31 - 40) for very severe RLS.
Brief Pittsburgh Sleep Quality Index (B-PSQI) | There will be three time points at which the measurement is assessed for both the study and the control group as follows: Pre-test: At the first day Post-test 1: two weeks later . Post-test 2: four weeks later.
  Brief Pittsburgh Sleep Quality Index (B-PSQI) is a self-reported measure with six components. The items are classified and evaluated in five categories: sleep quality, nocturnal awakenings, sleep efficiency, sleep duration, and sleep latency. Each sleep component is coded using a Likert scale ranging from 0 to 3. The sum of the five components gives a total score between 0 and 15, with higher values indicating poorer sleep quality. Scores from 0 to 5 indicate acceptable sleep quality, whereas scores of 6 or higher indicate poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Amjed A Shraida, PhD, Principal Investigator — Kufa University-Faculty of Nursing
Locations (1):
- Al-Sadder Medical City, Najaf, Al Kufa, Iraq

IPD SHARING:
Plan to Share IPD: No